CLINICAL TRIAL: NCT02704117
Title: Neurocircuitry of OCD: Effects Of Modulation
Brief Title: Neurocircuitry of Obsessive-Compulsive Disorder: Modulation by Transcranial Magnetic Stimulation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Butler Hospital (Other)
Collaborators: University of Rochester (Other); Harvard University (Other); University of Pittsburgh (Other); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P50MH106435 (NIH)
Record Dates: First submitted 2016-02-29; First posted 2016-03-09 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): Transcranial Magnetic Stimulation applied over the pre-supplementary motor area (pSMA), for ten sessions, Monday through Friday, over the course of two weeks.
  Interventions: Device: Transcranial Magentic Stimulation

INTERVENTIONS:
Device: Transcranial Magentic Stimulation — This is a form of mild brain stimulation delivered noninvasively. The device delivers pulses of magnetic energy through a coil placed on the scalp. The treatment takes 41 seconds, and takes place for ten sessions, Monday through Friday, over the course of two weeks
  Other Names: Continuous Theta Burst Stimulation (cTBS)

SUMMARY:
The purpose of this study is to test the effects of non-invasive neuromodulation, transcranial magnetic stimulation on brain function in individuals with obsessive-compulsive disorder (OCD). This study is focused on the mechanism(s) by which brain stimulation might change the functioning of regions implicated in OCD, and thereby inform possible future therapeutic uses.

ELIGIBILITY:
Inclusion Criteria:

* Current primary OCD diagnosis and current Y-BOCS total score of ≥16
* 18-70 years of age
* Ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent
* No use of psychiatric medications or stable psychiatric medication use for a minimum of 6 week prior to study entry
* Ongoing psychotherapy allowed if already established for three months or more before study entry

Exclusion Criteria:

* History of primary psychotic disorder or bipolar disorder
* Present acute suicidality
* History of head injury, epilepsy, or other clinically significant neurological illness except tic disorders
* Active systemic medical (metabolic, endocrine, chronic inflammatory, vascular, autoimmune) disease
* Premorbid intelligence quotient (IQ) estimate < 80
* Visual disturbance (<20/40 Snellen visual acuity, corrected)
* Current, or alcohol or illicit substance abuse/dependence in the last 3 months
* Contraindications to TMS or MRI: metallic foreign objects, e.g., aneurysm clips/pacemakers, or questionable history of metal fragments, claustrophobia
* Women who are pregnant or breastfeeding. All women participants of reproductive age are required to have a negative pregnancy test prior to enrollment and use medically acceptable birth control throughout the study (barrier and/or oral contraceptives)
* Current psychotic symptoms
* An increased risk of seizure, determined by history
* Medications judged to notably affect cortical excitability e.g., anticonvulsants or high-dose benzodiazepines (> 4 mg/day of clonazepam or equivalent)
* Predominant hoarding symptoms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2022-09 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in activation of pre-supplementary motor area/dorsal anterior cingulate cortex (pSMA/dACC) on functional magnetic resonance imaging (fMRI) during the Multi-Source Interference task (MSIT) | Baseline and 6 months

SECONDARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- See also: Related Info — https://butler.org/stim